CLINICAL TRIAL: NCT05427019
Title: Continuous Distal Adductor Canal Block With Periarticular Local Anesthetic Infiltration Versus Continuous Distal Adductor Canal Block Alone for Analgesia After Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 4-2022-0508
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Degenerative Osteoarthritis
MeSH Terms: conditions — Joint Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Distal adductor canal block (Active Comparator): Participants receiving continuous distal adductor canal block
  Interventions: Procedure: Distal adductor canal block
- Distal adductor canal block and Periarticular block (Active Comparator): Participants receiving continuous distal adductor canal block and periarticular block
  Interventions: Procedure: Distal adductor canal block and Periarticular block

INTERVENTIONS:
Procedure: Distal adductor canal block — All catheters were inserted under a full aseptic technique using a real-time ultrasound-guided in-plane approach by an experienced anesthesiologist. The adductor canal catheter is inserted 2cm above the adductor hiatus.
  Arms: Distal adductor canal block
Procedure: Distal adductor canal block and Periarticular block — All catheters were inserted under a full aseptic technique using a real-time ultrasound-guided in-plane approach by an experienced anesthesiologist. The adductor canal catheter is inserted 2cm above the adductor hiatus.The periarticular injection solution contained 20mL of 7.5 mg/mL ropivacaine, 30mg of ketorolac, and 0.3mL of 1.0 mg/mL epinephrine. These agents were mixed with normal saline to a combined volume of 50mL. The surgeon injected this mixture into the tensor fascia lata, subcutaneous tissues, abductors, short external rotators muscles, and structures in the capsule.
  Arms: Distal adductor canal block and Periarticular block

SUMMARY:
Continuous administration of local anesthetics to the distal adductor canal could spread into the popliteal fossa and contribute to analgesic effects on posterior knee pain. Periarticular local anesthetic infiltration is a component of multimodal joint pathways and the posterior knee capsule was among the tissues routinely infiltrated. It is expected that there will be overlapping effects of distal adductor canal block and periarticular injection. Therefore, we aim to compare the postoperative pain in the group that received only continuous distal adductor canal block and the group that received both continuous distal adductor canal block and periarticular injection. Sixty-six patients scheduled for total knee arthroplasty will be randomly divided into the two groups. In group 1, the adductor canal catheter is inserted 2cm above the adductor hiatus. In group 2, the adductor canal catheter is inserted where the nerve block performed in group 1 and periarticular injection are performed intraoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 19 years old or older, with American Society of Anesthesiologists Physical Status 1-3, and scheduled for elective unilateral total knee arthroplasty

Exclusion Criteria:

1. Allergy or intolerance to any of the drugs used in the study 2. Hepatic or renal insufficiency 3. Opioid dependency 4. Coagulopathy 5. Pre-existing neurologic or anatomic deficits in the lower extremities 6. Severe psychiatric illness

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-07-17 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Numeric rating scale pain score | postoperative 1 day morning (08:00-09:00 AM)
  Pain intensity at rest evaluated by an 11-point numeric rating scale (NRS: 0 = no pain, 10 = worst imaginable pain)

SECONDARY OUTCOMES:
Numeric rating scale pain score | postoperative 6 hours, postoperative 1 day afternoon (4:00-5:00 PM), postoperative 2 day morning (08:00-09:00 AM)
  Pain intensity at rest evaluated by an 11-point numeric rating scale (NRS: 0 = no pain, 10 = worst imaginable pain)

CONTACTS AND LOCATIONS:
Overall Officials: Yong Seon Choi, Principal Investigator — Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No